CLINICAL TRIAL: NCT00059137
Title: Respiratory Cycle Biofeedback During CT Guided Procedures
Brief Title: Breathing Cycle Biofeedback During Computed Tomography Procedures
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030166; 03-CC-0166
Record Dates: First submitted 2003-04-18; First posted 2003-04-18 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-03

CONDITIONS: Needle Biopsy; CAT Scan; X-Ray
Keywords: Gating; Respiratory Misregistration; Abdominal Belt; Percutaneous; CT Guided Biopsy; Respiratory Cycle; Needle Biopsy

SUMMARY:
This study will evaluate the effectiveness of a flexible belt device in guiding patient breathing during computed tomography (CT)-guided needle biopsy. When patients undergo CT scanning to help guide the physician during a tissue biopsy, they are usually asked to hold their breath while the scan is taken of certain parts of the body. When the first scan is completed, the patients are allowed to breathe, and are then asked to hold their breath again while the needle is advanced towards the tissue to be biopsied. Since body organs and tissues move with breathing, this study will try to stop the patient's breathing at the same place in the breathing cycle to ensure that the biopsy target stays still and in the same place. This study will see if the flexible belt, used with a computer screen that charts the patient's breathing, will improve the patient's ability to stop breathing at the same place in the breathing cycle before and during the biopsy.

Patients 18 years of age and older who have a lesion requiring a needle biopsy in the chest or abdominal area may be eligible for this study. The biopsy procedure must require CT scan guidance.

Participants will undergo the following procedures:

* Breathing exercise: A flexible, loose-fitting belt is placed around the patient's abdomen and the patient is asked to stop breathing in the following ways: 1) take a deep breath in and hold; 2) breathe deeply out and hold; and 3) breathe regularly and hold.
* Needle biopsy: The patient is positioned in a CT scanner and is asked to hold his or her breath while an initial scan is taken. Then the patient is taken out of the scanner and the place the needle entry site for the biopsy is marked on the skin. A local anesthetic is applied to the site and the patient is asked to hold his or her breath the same way as before. During this breath hold, the patient may or may not be shown a computer screen displaying a graph of the patient's breathing and the point in the cycle of the previous breath hold. The biopsy is then performed with CT guidance. While the CT pictures are being taken, the patient is again asked to breathe and hold his or her breath as before. When the biopsy is completed, the belt device is removed.

DETAILED DESCRIPTION:
This study will examine the use of a flexible belt placed across the patient's abdomen to sense and plot the patient's respiratory cycle. The point in the respiratory cycle at which the patient holds his/her breath will be recorded at different levels and correlated with CT scans and prior patient breathing levels. Our hypothesis is that a graphical representation of the respiratory cycle may make it easier for the patient to hold his or her breath at the same level each time a CT scan is obtained, or a needle is inserted. If this is true, then this should translate into faster safer procedures, with potentially less ionizing radiation, although this endpoint is not defined in this particular study.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients must fulfill all of the following criteria to be eligible for study admission:

1. All patients must have a lesion needing biopsy in the chest or abdominal areas in special procedures requiring CT scan guidance.
2. age greater than 18 years.
3. No serious concurrent medical illness that would preclude the patient from making a rational informed decision on participation.
4. The ability to understand and willingness to sign a written informed consent form, and to comply with the protocol. If in question, an ethics consult will be obtained.

EXCLUSION CRITERIA:

Patients with any of the following will be excluded from study entry:

1. Patients with an altered mental status that precludes understanding or consenting for the biopsy procedure will be excluded from this study.
2. patients unable to hold breath for more than 5 seconds.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2003-04; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Tomiyama N, Mihara N, Maeda M, Johkoh T, Kozuka T, Honda O, Hamada S, Yoshida S, Nakamura H. CT-guided needle biopsy of small pulmonary nodules: value of respiratory gating. Radiology. 2000 Dec;217(3):907-10. doi: 10.1148/radiology.217.3.r00dc10907. PMID 11110962
- [Background] Frohlich H, Dohring W. A simple device for breath-level monitoring during CT. Radiology. 1985 Jul;156(1):235. doi: 10.1148/radiology.156.1.4001413.
- [Background] Connolly BL, Chait PG, Duncan DS, Taylor G. CT-guided percutaneous needle biopsy of small lung nodules in children. Pediatr Radiol. 1999 May;29(5):342-6. doi: 10.1007/s002470050603. PMID 10382211